CLINICAL TRIAL: NCT00733343
Title: Treatment of Sleep-Disordered Breathing With Predominant Central Sleep Apnea by Adaptive Servo Ventilation in Patients With Heart Failure
Brief Title: Treatment of Predominant Central Sleep Apnoea by Adaptive Servo Ventilation in Patients With Heart Failure
Acronym: Serve-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: CRI-The Clinical Research Institute GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01; ISRCTN19572887 (Other: International Standard Randomised Controlled Trials)
Record Dates: First submitted 2008-02-14; First posted 2008-08-13 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure; Sleep Disordered Breathing
Keywords: heart failure (HF); sleep disordered breathing (SDB); sleep apnea; left ventricular systolic dysfunction
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes; Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Active Comparator): treatment with Adaptive Servoventilation (Europe: AutoSet CS (USA: VPAP (Variable Positive Airway Pressure) Adapt SV)) + standard medical therapy according to applicable guidelines (ESC, ACC/AHA)
  Interventions: Device: Europe: AutoSet CS (USA: VPAP Adapt SV)
- Control Group (No Intervention): standard medical therapy according to applicable guidelines (ESC, ACC/AHA)

INTERVENTIONS:
Device: Europe: AutoSet CS (USA: VPAP Adapt SV) — At least 3 hours average daily usage time
  Arms: Treatment Group

SUMMARY:
The purpose of this trial is to evaluate the long-term effects and cost-effectiveness of adaptive servo-ventilation (ASV) on the mortality and morbidity of patients with stable heart failure due to left ventricular systolic dysfunction, already receiving optimal medical therapy, who have sleep disordered breathing (SDB) that is predominantly central sleep apnea. Assumptions: the intervention reduces the hazard rate by 20%. The event rate in the control group is 35% in the first year. It is assumed that the hazard rate is constant over time.

DETAILED DESCRIPTION:
Objective: The purpose of this trial is to evaluate the long-term effects and cost-effectiveness of adaptive servo-ventilation (ASV) on the mortality and morbidity of patients with stable heart failure due to left ventricular systolic dysfunction, already receiving optimal medical therapy, who have sleep disordered breathing (SDB) that is predominantly central sleep apnea.

Study Design: Randomized, multicentre, international trial with parallel group design, with patients randomized to either control (optimal medical management) or active treatment (optimal medical treatment plus use of adaptive servoventilation) in a 1:1 ratio. There will be no sham-positive airway pressure treatment in the control arm. Assumptions: the intervention reduces the hazard rate by 20%. The event rate in the control group is 35% in the first year. It is assumed that the hazard rate is constant over time. The trial is an event driven design: the final analysis is to be performed latest when 651 events have been observed. The primary analysis is in the intention-to-treat population that consists of all patients randomized.

Number of Patients: 1116 patients will be randomly assigned to one of the two treatment groups. A 20% drop out rate is estimated.

Selection criteria: Patients at the age of or over 22 years with severe chronic heart failure (chronic HF), New York Heart Association (NYHA) class III-IV or NYHA class II with at least one hospitalization for HF within the last 24 months, with Left Ventricular Ejection Fraction (LVEF) less or equal 45% by means of echocardiography, radionuclide ventriculography or cardiac MRI and Sleep Disordered Breathing (SDB) (apnoea-hypopnoea-index (AHI > 15/h) with 50% central events and a central AHI ≥ 10/h, no change of medication and no hospitalization for more than 1 month before randomization and medical therapy according to the applicable guidelines (European Society of Cardiology (ESC) and American College of Cardiology/American Heart Association (ACC/AHA) respectively).

Primary Endpoints: Time to first event of:

1. all cause mortality or unplanned hospitalisation/prolongation of hospitalisation for worsening heart failure
2. cardiovascular mortality or unplanned hospitalisation/prolongation of hospitalisation for worsening heart failure.
3. all cause mortality or all cause unplanned hospitalisation/prolongation of hospitalisation Heart transplantation, appropriate shock from implantable cardioverter-defibrillator (ICD), long term assist device (LTAD) insertion and survived resuscitation of sudden cardiac arrest are counted as cardiovascular death, survived resuscitation for other reasons is counted as all cause death.

The three combinations are not tested in parallel but in this hierarchical order.

Secondary Endpoints : Time until death, non cardiovascular death, cardiovascular death, hospitalization due to deterioration of heart failure or cardiovascular death, hospitalization for other reasons or death, hospitalization for cardiovascular cause or cardiovascular death, percent of follow-up (FU) days which patient survives and is not hospitalized for cardiovascular cause, percent of follow up days which patient survives and is not hospitalized for other reason, time to first adequate shock (in patients with ICD, evaluation of appropriateness will also be made by the ERC) or cardiovascular death, changes in NYHA class as compared to baseline, changes in difference in health costs between the two treatment groups, changes in QoL (Minnesota, Euroqol 5D (EQ5D)) as compared to baseline, changes in renal function (based on serum creatinine) as compared to baseline, changes in result of Six Minute Walking Test (6MWT) (50) as compared to baseline,changes of AHI and oxygen desaturation index compared to baseline, AHI below 10 per hour at twelve months and Oxygen desaturation index (ODI) below 5 per hour at twelve months, atrial fibrillation at follow-up visits.

Number and cost of hospitalizations (with tariff/diagnostic-related Group (DRG), diagnoses and procedures for calculating DRG or length of stay and level of care provided), cost of care (technology and service, nursing, physicians visit) related to ventilation, difference in utilities / QoL (Minnesota and EQ5D) compared to control arm, difference in cost of resources consumed, cost-efficacy, cost-utility. Secondary target parameters will be measured at the last follow up or at the last available observation within FU.

Scheduled follow up : Minimum follow up time will be 24 months, maximum about 70 months. There will be a final assessment for each patient at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 22 years old
* Chronic heart failure (at least 12 weeks since diagnosis) according to the current applicable guidelines (ESC, ACC/AHA)
* Left ventricular systolic dysfunction (LVEF ≤45% by imaging method such as echocardiography, radionuclide angiography, left ventriculography, or cardiac magnetic resonance imaging) documented less than 12 weeks before randomisation
* NYHA class III or IV at the time of inclusion or NYHA class II with at least one hospitalisation for HF in the last 24 months
* No hospitalisation for heart failure for at least 4 weeks prior to inclusion
* Optimised medical treatment according to applicable guidelines with no new class of disease modifying drug for more than 4 weeks prior to randomisation. In case of no beta blockers or ACE (angiotensin converting Enzyme) inhibitors/ ARB (angiotensin receptor blocker) antagonists the reasons must be documented
* SDB (AHI > 15/h with ≥ 50% central events and a central AHI ≥ 10/h, derived from polygraphy or polysomnography (based on total recording time (TRT)), documented less than 4 weeks before randomisation. Flow measurement has to be performed with nasal cannula
* Patients for whom the use of AutoSet CS2 (TM)/VPAP Adapt may be contra-indicated because of symptomatic hypotension or significant intravascular volume depletion or pneumothorax or pneumomediastinum
* Patient is able to fully understand study information and signed informed consent

Exclusion Criteria:

* Significant COPD (chronic obstructive pulmonary disease) with Forced Expiratory Volume within one second (FEV1) <50% (European Respiratory Society criteria) in the last four weeks before randomisation
* Oxygen saturation at rest during the day ≤ 90% at inclusion
* Current use of Positive Airway Pressure (PAP) - therapy
* Life expectancy < 1 year for diseases unrelated to chronic HF
* Cardiac surgery, Percutaneous coronary intervention (PCI), Myocardial Infarction (MI) or unstable angina within 6 months prior to randomisation
* CRT (cardiac resynchronisation therapy)-implantation or ICD-implantation scheduled or within 6 months prior to randomisation
* Transient ischemic attack (TIA) or Stroke within 3 months prior to randomisation
* Primary hemodynamically significant uncorrected valvular heart disease, obstructive or regurgitant, or any valvular disease expected to lead to surgery during the trial
* Acute myocarditis/pericarditis within 6 months prior to randomisation
* Untreated or therapy refractory Restless legs-Syndrome (RLS) according to criteria listed in Appendix IX at the time of study entry
* Pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1325 (Actual)
Dates: Start 2008-02; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Teschler, Prof., Principal Investigator — Universitätsklinikum Essen; Martin Cowie, Prof., Principal Investigator — National Heart and Lung Institute (NHLI) Brompton Hospital, London
Locations (266):
- Australia (6):
  - Westmead Hospital, Westmead, New South Wales
  - Rivercity Private Hospital, Auchenflower, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincents and Mercy Private Hospital, Melbourne, Victoria
  - Melbourne Sleep Disorders Centre, East Melbourne, Victoria 3002
  - Hollywood Private Hospital (CVS), Nedlands, Western Australia
- St. Anne's University Hospital BRNO, Brno, Czechia
- Denmark (6):
  - Århus Universitets Hospital, Århus C
  - Århus Universitets Hospital Skejby, Århus N
  - Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Dansk Center For Søvnmedicin, Glostrup Municipality
  - Glostrup Hospital, Glostrup Municipality
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Unesta Research Centre, Tampere
  - Tampere University Hospital, Pirkanmaa sairaanhoitopiiri, Tampere
- France (49):
  - Cardiologist Dr. Papola, Amnéville
  - CHU Angers, Angers
  - Centre Hospitalier d'Antibes Juan-les-Pins, Antibes
  - Hopital Prive d'Antony, Antony
  - CH Belfort, Belfort
  - CH de Besancon, Besançon
  - Centre Hospitalier de Béziers, Béziers
  - Clinique du Tondu, Bordeaux
  - Hôpital St. André, Bordeaux
  - Praxis Cardiologique Dr. Puel, Bordeaux
  - Praxis Cardiologique Dr. Wickers, Bordeaux
  - CHU Bordeaux, Hopital Pellegrin, Bordeaux
  - CHU de Caen, Caen
  - Centre Hospitalier de Cannes, Cannes
  - Hopital Henri Mondor, Créteil
  - Hôpital Sud, Échirolles
  - CH de Forbach, Hospitalor, Hopital Marie Madeleine-Pneumology, Forbach
  - CH de Forbach-Cardiology, Forbach
  - Clinique Mutualiste des Eaux Claires, Grenoble
  - CHU Grenoble, Hopital Michallon, Grenoble
  - CH Haguenau, Haguenau
  - Clinique de L'Union, L'Union
  - CHU Lille- Hopital Cardiologique, Lille
  - CHU Lille-Sleep medicine, Lille
  - Polyclinique La Louviere, Lille
  - Hospices Civils de Lyon, Hopital de la Croix-Rousse, Lyon
  - CHR Metz, Hôpital de Bon-Secours, Metz
  - CH Montbeliard, Montbéliard
  - CHU de Montpellier, Montpellier
  - CH Intercommunal André Grégoire, Montreuil
  - CH de Mulhouse, Hopital Emile Muller, Mulhouse
  - Clinique les Fleurs, Ollioules
  - Hôpital Bichat, Paris
  - CHU Tenon, Paris
  - CHU de Bordeaux, Hopital Haut Leveque, Pessac
  - CHU de Poitiers, Poitiers
  - Cabinet de cardiologie, Pont-à-Mousson
  - CH Rene Dubos, Pontoise
  - Polyclinique Saint-Laurent, Rennes
  - CHU de Rouen, Hopital de Bois Guillaume, Rouen
  - CH Lemire - St Avold, Saint-Avold
  - CH de St Dié des Vosges, Saint-Dié
  - CHU de Saint-Etienne, Hopital Nord, Saint-Etienne
  - Clinique des Trois Frontières, Saint-Louis
  - CHU Toulouse, Hopital de Rangueil, Toulouse
  - CHU Toulouse, Hopital Larrey, Toulouse
  - CH Trouville, Trouville
  - CHU de Nancy, Hopital Brabois, Vandœuvre-lès-Nancy
  - Ch St. Nicolas, Verdun
- Germany (185):
  - Cardiopraxis Ingelheim, Ingelheim, Rhineland-Palatinate
  - Praxis Dr. Frieske, Aachen
  - Universitätsklinikum Aachen, Aachen
  - DRK Krankenhaus, Alzey
  - Gemeinschaftspraxis Weiß / Dr. Heesing, Arnsberg
  - Zentralklinikum Bad Berka, Bad Berka
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Klinik Lazariterhof, Bad Krozingen
  - Schlaflabor Breisgau, Bad Krozingen
  - Praxis Dr. Bauer, Bad Mergentheim
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Oberlausitz-Kliniken gGmbH, Bautzen
  - Kardiologie Brühl, Bergheim
  - Kardiopraxis Rheinberg, Bergisch Gladbach
  - Charité Campus Mitte - Kardiologie, Berlin
  - Charité Campus Mitte CCM- Schlafmedizinisches Zentrum, Berlin
  - POLIKUM Friedenau, Berlin
  - Gemeinschaftspraxis Groß-Ziethener Chaussee, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Evangelische Lungenfachklinik Buch, Berlin
  - Jüdisches Krankenhaus Berlin, Berlin
  - Charité Campus Virchow Klinikum, Berlin
  - Praxis Westend, Berlin
  - Herzzentrum Brandenburg, Bernau
  - Praxis für Lunge, Herz und Schlaf, Bielefeld
  - Kardiologie Gemeinschaftspraxis Dres Tenholt&Metzger&Dexling, Bochum
  - Universitätsklinikum Bergmannsheil, Bochum
  - Augusta Krankenanstalten Bochum, Bochum
  - St.-Josephs-Hospital, Bochum
  - Kardiologie Kemnade, Bochum
  - Kardiologische Praxis Dr. Staubach, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Kardiologische Praxis Marschner, Bonn
  - Helios Klinikum Borna, Borna
  - Gemeinschaftspraxis Kardiologie, Bottrop
  - Klinikum Bremen Ost, Bremen
  - Kardiologie Brühl, Brühl
  - Mediclin Rehazentrum Spreewald, Burg
  - Gemeinschaftspraxis Kardiologie Dr. Becker, Castrop-Rauxel
  - Kardiologische Praxis Dr. Isbruch, Castrop-Rauxel
  - MVZ am Küchwald, Chemnitz
  - Klinikum Coburg GmbH, Coburg
  - St.-Vinzenz Hospital, Cologne
  - Kardiologische Praxis Dr. Fritsch, Cologne
  - Malteser Krankenhaus St.Hildegardis, Cologne
  - Prof. Franzen Institut, Cologne
  - Praxis Dr. Anselm Bäumer, Cologne
  - Gemeinschaftspraxis Dres. Gysan/Heinzler/May, Cologne
  - Fachkrankenhaus Coswig, Coswig
  - Carl-Thiem-Klinikum gGmbH, Cottbus
  - Ambulantes Zentrum für Lungenkrankheiten&Schlafmedizin, Cottbus
  - MECS Cottbus GmbH, Cottbus
  - Praxis Dr. Hecker, Dortmund
  - Kardiologische Praxis Dr. Golling, Dortmund
  - Clinical Trial Site Services, Dortmund
  - Kardiologische Praxis Dr. Wetzel, Dortmund
  - Kardiologische Praxis Dr. Lodde, Dortmund
  - Kardiologische Praxis Dr. Dröse, Dortmund
  - Facharztzentrum Dresden-Neustadt GbR, Dresden
  - Gemeinschaftspraxis Dres. Schmidt/Gronke, Dresden
  - Praxis Dr. Hohensee, Dresden
  - Herzzentrum Universität Dresden, Dresden
  - goMedus Gesundheitszentrum, Düsseldorf
  - Kardiologische Praxis Dr. Horowitz, Düsseldorf
  - Evangelisches Krankenhaus, Düsseldorf
  - Kardiologische Praxis Dr. Raff, Düsseldorf
  - Florence-Nightingale Krankenhaus, Düsseldorf
  - Kardiologie Oberkassel, Düsseldorf
  - Gemeinschaftspraxis PD. Dr. Lankisch, Düsseldorf
  - Fachärzte für Innere Medizin Dres Ritter, Richter, Mehrer, Kahl, Emmendingen
  - Helios Klinikum Erfurt-Kardiologie, Erfurt
  - Helios Klinikum Erfurt-Schlafmedizin, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Westdeutsches Herzzentrum, Universitätsklinikum Essen, Essen
  - Kardiologische Praxis Dr. Cord Müller, Essen
  - Schwerpunktpraxis Kardiologie Drs. Ophoff/Fritzsch, Essen
  - Kardiologische Praxis Prof. Winter, Essen
  - Kardiologie Praxis Dr. Bonnekamp, Essen
  - Praxis Dr. Tekiyeh, Essen
  - Elisabeth-Krankenhaus Essen, Essen
  - Ruhrlandklinik Essen, Essen
  - Praxis Dr. Rau, Essen
  - Kath. Kliniken Essen / Philippusstift, Essen
  - Gemeinschaftspraxis Dres. Guckenbiehl, Flonheim
  - Kardiologische Praxis Dr. Kruse, Forst
  - CardioVasculäres Centrum Frankfurt, Frankfurt
  - Praxis Dr. Diedrichs, Frechen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Gemeinschaftspraxis Dres. Böhmeke/Schmidt, Gladbeck
  - Kardiologische Praxis Dr. Hug, Günzburg
  - Kardiologische Praxis Gütersloh, Gütersloh
  - Gemeinschaftspraxis Dres Leischik/Littwitz, Hagen
  - Kardiologische Praxis Dr. Arens, Hagen
  - Gemeinschaftspraxis Dres. Subin/Lutter, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Internistenpraxis Alstertal Hamburg, Hamburg
  - Kardiologische Praxis Dr. Cierpka, Hanover
  - Praxis Dr. Hötte, Hanover
  - Siloah Krankenhaus, Hanover
  - Kardiologische Praxis Dr. Hartung, Hanover
  - MH Hannover, Hanover
  - Klinikum Hannover Oststadt-Heidehaus, Hanover
  - Praxis Dr. Durak, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Kardiologische Praxis Dr. Furche, Herne
  - Gemeinschaftspraxis Dr. Bruch, Herne
  - Kardiologische Praxis Dr. Schlichting, Herne
  - Augusta-Kranken-Anstalt gGmbH Thoraxzentrum Ruhrgebiet, Herne
  - St. Elisabeth-Hospital Herten gGmbH, Herten
  - Lungenfachklinik Immenhausen, Immenhausen
  - Gemeinschaftspraxis Dres. Dobler/Turin, Karlstadt am Main
  - Ambulantes Herzzentrum Kassel, Kassel
  - Kardiologische Praxis Dr. Siegfried Frickel, Kempen
  - Klinikum Dahme-Spreewald GmbH, Königs Wusterhausen
  - Praxis Dr. Krater, Krefeld
  - Helios Klinikum Krefeld, Krefeld
  - Universitätsklinikum Leipzig-Herzzentrum, Leipzig
  - Helios Krankenhaus Leisnig, Leisnig
  - Gemeinschaftspraxis Dr. Hilgedieck/Sava, Lengerich
  - Kardiologische Praxis Dr. Faber, Lindlar
  - Ärztezentrum Holthausen-Biene, Lingen
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck-Kardiologie, Lübeck
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck-Schlaflabor, Lübeck
  - Klinikum der Johannes Gutenberg-Universität Mainz, Mainz
  - Cardiopraxis Ingelheim, Mainz
  - Universitätsklinikum Mannheim-Schlafmedizin, Mannheim
  - Gemeinschaftspraxis Dres. Heifer/Loster/Schernus, Mannheim
  - Gemeinschaftspraxis für Herz & Gefäße, Mannheim
  - Universitätsklinik Mannheim-Kardiologie, Mannheim
  - Gemeinschaftspraxis Dres. Brandt / Jakobs, Mannheim
  - Universitätsklinikum Gießen / Marburg, Standort Marburg-Schlafmedizin, Marburg
  - Universitätsklinikum Gießen/Marburg Standort Marburg-Kardiologie, Marburg
  - Praxis Dr. Schnabel, Meissen
  - Gemeinschaftspraxis Dr. Jocham, Memmingen
  - Praxis Für Kardiologie Dr. med. Menz, Menden
  - Krankenhaus Bethanien, Moers
  - Kardiologische Praxis Dr. Schön, Mühldorf
  - Evangelisches Krankenhaus Mülheim, Mülheim
  - Kardiologie am Rotkreuzplatz, München
  - Lungenärzte am Rotkreuzplatz, München
  - Gemeinschaftspraxis Dres. Wauer / Windstetter, München
  - Kardiologische Praxis Dr. Herholz, München
  - Klinik Augustinum München, München
  - Praxis Dres. Böhme/Linke, München
  - Kardiologische Praxis Dr. Muradi, Münster
  - Universitätsklinikum Münster, Münster
  - Praxis für Kardiologie Dr. med. Hewing, Münster
  - Lukaskrankenhaus GmbH, Neuss
  - Kardiologische Praxis Nienburg, Nienburg
  - Klinikum Nürnberg Nord, Nuremberg
  - Klinikum Nürnberg Süd, Nuremberg
  - Kardiologische Praxis Dr. Gumbrecht, Ochtrup
  - Kardiologische Praxis Dr. Wiethölter, Radebeul
  - Praxis für Kardiologie Ratingen, Ratingen
  - Praxis Dr. Fröhlich, Ratingen
  - DRK Krankenhaus Mölln-Ratzeburg, Ratzeburg
  - Ambulantes Cardiovaskuläres Centrum, Ravensburg
  - Gemeinschaftspraxis Dr. Weber/Dr. Feja, Recklinghausen
  - Knappschafts-Krankenhaus Recklinghausen, Recklinghausen
  - Universitätsklinikum Regensburg, Regensburg
  - Krankenhaus Reinbek St. Adolf-Stift, Reinbek
  - Praxis Dr. Hein, Reinbek
  - Praxis Dr. Nebel, Rheine
  - Praxis Dr. Kestermann, Rheine
  - Praxis Dr. Ebeling, Schönefeld
  - Kardiologische Praxis Dr. Heinze, Schwerte
  - Praxisgemeinschaft Cardio-Soest, Soest
  - Facharztzentrum Sonneberg, Sonneberg
  - Kreiskrankenhaus Stollberg GmbH, Stollberg
  - Klinikum Uelzen GmbH, Uelzen
  - Herzklinik Ulm Dr. Haerer und Partner, Ulm
  - Zentrum für Innere Medizin Uni Ulm, Ulm
  - Katharinen Hospital Unna, Unna
  - Kardiologische Praxis Dr. Burkhard-Meier, Viersen
  - Praxis Dr. Gerritsen, Waldkraiburg
  - Fachkliniken Wangen, Wangen
  - Stiftungsklinik Weißenhorn, Weißenhorn
  - Kardiologische Praxis Dr. Vrettos, Witten
  - Kardiologische Praxis Dr. Rudolf/ Dr. Bernhardt, Worms
  - Missionsärztliche Klinik Würzburg, Würzburg
  - Universitätsklinikum Würzburg, Würzburg
  - Evangel. Khs Zweibrücken, Zweibrücken
- University Medical Center Groningen, Groningen, Netherlands
- Norway (3):
  - Ullevål University Hospital, Oslo
  - Oslo University Hospital, Rikshospitalet, Oslo
  - Stavanger AS, Stavanger
- Sweden (4):
  - Sahlgrenska University Hospital / Östra, Gothenburg
  - Specialistläkarmottagning Residenset AB, Jönköping
  - Skaraborgs Hospital, Lidköping
  - Linköping University Hospital, Linköping
- Switzerland (2):
  - Cardiocentro Ticino, Lugano
  - Ospedale Regionale di Lugano, Lugano
- United Kingdom (6):
  - Castle Hill Hospital, Cottingham, East Yorkshire
  - Chesterfield Royal Hospital, Chesterfield
  - Brompton Hospital, London
  - Freeman Hospital, Newcastle
  - Musgrove Park Hospital, Taunton
  - Royal Wolverhampton Hospitals NHS Trust, Wolverhampton

REFERENCES:
- [Result] Cowie MR, Wegscheider K, Teschler H. Adaptive Servo-Ventilation for Central Sleep Apnea in Heart Failure. N Engl J Med. 2016 Feb 18;374(7):690-1. doi: 10.1056/NEJMc1515007. No abstract available. PMID 26886528
- [Result] Eulenburg C, Wegscheider K, Woehrle H, Angermann C, d'Ortho MP, Erdmann E, Levy P, Simonds AK, Somers VK, Zannad F, Teschler H, Cowie MR. Mechanisms underlying increased mortality risk in patients with heart failure and reduced ejection fraction randomly assigned to adaptive servoventilation in the SERVE-HF study: results of a secondary multistate modelling analysis. Lancet Respir Med. 2016 Nov;4(11):873-881. doi: 10.1016/S2213-2600(16)30244-2. Epub 2016 Aug 31. PMID 27592224
- [Result] Woehrle H, Cowie MR, Eulenburg C, Suling A, Angermann C, d'Ortho MP, Erdmann E, Levy P, Simonds AK, Somers VK, Zannad F, Teschler H, Wegscheider K. Adaptive servo ventilation for central sleep apnoea in heart failure: SERVE-HF on-treatment analysis. Eur Respir J. 2017 Aug 31;50(2):1601692. doi: 10.1183/13993003.01692-2016. Print 2017 Aug. PMID 28860264
- [Derived] Tamisier R, Pepin JL, Woehrle H, Salvat M, Barone-Rochette G, Rocca C, Vettorazzi E, Teschler H, Cowie M, Levy P. Effect of adaptive servo-ventilation for central sleep apnoea in systolic heart failure on muscle sympathetic nerve activity: a SERVE-HF randomised ancillary study. Eur Respir J. 2023 Feb 9;61(2):2200384. doi: 10.1183/13993003.00384-2022. Print 2023 Feb. PMID 36229051
- [Derived] Shafazand S, Badr MS. Adaptive Servo-Ventilation and Central Apnea Associated with Systolic Heart Failure. J Clin Sleep Med. 2016 Jan;12(1):147-50. doi: 10.5664/jcsm.5420. No abstract available. PMID 26888594
- [Derived] Cowie MR, Woehrle H, Wegscheider K, Angermann C, d'Ortho MP, Erdmann E, Levy P, Simonds AK, Somers VK, Zannad F, Teschler H. Adaptive Servo-Ventilation for Central Sleep Apnea in Systolic Heart Failure. N Engl J Med. 2015 Sep 17;373(12):1095-105. doi: 10.1056/NEJMoa1506459. Epub 2015 Sep 1. PMID 26323938

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: treatment with Adaptive Servoventilation (Europe: AutoSet CS (USA: VPAP Adapt SV)) + standard medical therapy according to applicable guidelines (ESC, ACC-american college of cardiology/AHA)
  Europe: AutoSet CS (USA: VPAP Adapt SV): At least 3 hours average daily usage time
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 666 | 659
Completed | 583 | 578
Not Completed | 83 | 81

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: treatment with Adaptive Servoventilation (Europe: AutoSet CS (USA: VPAP Adapt SV)) + standard medical therapy according to applicable guidelines (ESC, ACC/AHA)
  Europe: AutoSet CS (USA: VPAP Adapt SV): At least 3 hours average daily usage time
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 666 | 659 | 1325
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (9.5) | 69.3 (10.4) | 69.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 60 | 127
  Male | 599 | 599 | 1198
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 3 | 4 | 7
  Netherlands | 0 | 1 | 1
  Sweden | 20 | 19 | 39
  Norway | 5 | 5 | 10
  Finland | 4 | 3 | 7
  Denmark | 12 | 12 | 24
  United Kingdom | 18 | 19 | 37
  Australia | 16 | 13 | 29
  France | 119 | 123 | 242
  Switzerland | 2 | 1 | 3
  Germany | 467 | 459 | 926
NYHA class [Count of Participants; unit: Participants] — New York Heart Association (NYHA). Class I: No Limitation of physical activity. [...] Class II: Slight Limitation of physical activity. Comfortable at rest, but less than ordinary physical activity results in undue breathlessness, fatigue, or palpitations. Class III: Marked Limitation of physical activity. Comfortable at rest, but less than ordinary physical activity results in [...].Class IV: Unable to carry on any physical activity without discomfort. Symptoms at rest can be present. If any physical act is undertaken, discomfort is increased. Ref.: ESC Guidelines 2016 (c) ESC 2016
  Participants
    NYHA II | 195 | 194 | 389
    NYHA III | 456 | 454 | 910
    NYHA IV | 11 | 6 | 17
    not assessed | 4 | 5 | 9
Diabetes [Count of Participants; unit: Participants] | 254 | 252 | 506
Cause of Heart Failure [Count of Participants; unit: Participants]
  ischemic | 390 | 366 | 756
  nonischemic | 263 | 276 | 539
  not assessed | 13 | 17 | 30
Electrocardiographic Finding [Count of Participants; unit: Participants]
  sinus rhythm | 372 | 395 | 767
  atrial fibrillation | 178 | 147 | 325
  other | 100 | 104 | 204
  not assessed | 16 | 13 | 29
Implanted device [Count of Participants; unit: Participants]
  no device | 304 | 295 | 599
  non-CRT(cardiacresynchronisation therapy)pacemaker | 32 | 29 | 61
  ICD (implantable cardioverter defibrillator) | 163 | 161 | 324
  CRT-P | 14 | 21 | 35
  CRT-D | 153 | 153 | 306
Concomitant cardiac medication [Count of Participants; unit: Participants] — Population: The values count the number of patients who have taken the respective medication.
  Participants
    ACE inhibitor or ARB(AT1 recept blocker) | 613 | 603 | 1216
    beta-blocker | 612 | 611 | 1223
    aldosterone antagonist | 316 | 325 | 641
    diuretic | 561 | 561 | 1122
    cardiac glycoside: number analyzed (Participants) | 666 | 657 | 1323
    cardiac glycoside | 149 | 124 | 273
    antiarrhythmic drug | 128 | 89 | 217

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality or Unplanned Hospitalisation/Prolongation of Hospitalisation for Worsening Heart Failure
Time Frame: time to first event, assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 360 | 335

2. Primary Outcome: Cardiovascular Mortality or Unplanned Hospitalisation/Prolongation of Hospitalisation for Worsening Heart Failure
Time Frame: time to first event, assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 345 | 317

3. Primary Outcome: All Cause Mortality or All Cause Unplanned Hospitalisation/Prolongation of Hospitalisation
Time Frame: time to first event, assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 482 | 465

4. Secondary Outcome: Death From Any Cause
Time Frame: the last follow up or at the last available observation within Follow Up (FU), assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 232 | 193

5. Secondary Outcome: Non-cardiovascular Death
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 33 | 35

6. Secondary Outcome: Cardiovascular Death
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 199 | 158

7. Secondary Outcome: Unplanned Hospitalisation/Prolongation of Hospitalisation Due to Worsening of Heart Failure
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 287 | 272

8. Secondary Outcome: Unplanned Hospitalisation/Prolongation of Hospitalisation for Other Reasons or Death
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 452 | 448

9. Secondary Outcome: Adequate Shock in Patients With ICD (Evaluation of Appropriateness Will Also be Made by the Endpoint Review Committee, ERC), Long-Term Atrial Defibrillator Insertion or Cardiovascular Death
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 45 | 65

10. Secondary Outcome: First Survived Resuscitation for Any Reason (Evaluation Will Also be Made by the ERC)
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 25 | 19

11. Secondary Outcome: First Survived Resuscitation of Sudden Cardiac Arrest (Evaluation Will Also be Made by the ERC)
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Participants | 18 | 16

12. Secondary Outcome: Age Baseline
Time Frame: 1 x at Baseline
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
years | 69.6 (9.5) | 69.3 (10.4)

13. Secondary Outcome: Body Weight Baseline
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
kg | 85.6 (15.8) | 86.1 (17.5)

14. Secondary Outcome: Body Mass Index (BMI) Baseline
Time Frame: 1 x baseline
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
kg/cm2 | 28.4 (4.7) | 28.6 (5.1)

15. Secondary Outcome: Left Ventricular Ejection Fraction at Baseline
Time Frame: 1x at baseline
Measure: Mean (Standard Deviation); unit: %total vol ventricle
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
%total vol ventricle | 32.2 (7.9) | 32.5 (8.0)

16. Secondary Outcome: Blood Pressure Systolic Baseline
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
mm Hg | 122.3 (19.0) | 122.1 (19.6)

17. Secondary Outcome: Blood Pressure Diastolic Baseline
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
mm Hg | 73.7 (11.3) | 73.3 (11.5)

18. Secondary Outcome: Hemoglobine Baseline
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
g/dl | 13.8 (1.6) | 13.9 (1.5)

19. Secondary Outcome: Creatinine Baseline
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
mg/dl | 1.4 (0.6) | 1.4 (0.6)

20. Secondary Outcome: Glomerular Filtration Rate Baseline
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
ml/min/1.73m2 | 57.8 (21.1) | 59.3 (20.8)

21. Secondary Outcome: 6-Min Walk Distance
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
m | 334.0 (126.4) | 337.9 (127.5)

22. Secondary Outcome: Epworth Sleepiness Scale (ESS)
Description: Measure Description: ESS is a self-administered questionnaire. It contains 8 questions. Questions are rated on a 4-point Likert scale (0-3); 0= would never doze, 3=high Chance of dozing. Range of scores 0-24. Global score= sum of all item scores. Copyright (c)MW Johns
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: total score ESS
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
total score ESS | 7.0 (4.3) | 7.1 (4.6)

23. Secondary Outcome: Apnoea-Hypopnea-Index (AHI) at Baseline
Description: Measure Description: The AHI is an index to describe the severity of Sleep Apnea. Apnea is cessation of breathing during sleep. Hypopnea is diminished breathing during sleep. The number of Apneas and Hypopneas are added up and divided by hours of sleep (Apneas + Hypopneas per hour). An AHI ranging from 5-15 describes mild Sleep Apnea. AHI 15-30 describes moderate Sleep Apnea. AHI >30 describes severe Sleep Apnea.
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
events/hour | 31.2 (12.7) | 31.7 (13.2)

24. Secondary Outcome: Central Apnoea Index/Total AHI
Description: Measure Description: Central apneas are partial or complete cessations of airflow caused by reduced or stopped neural Stimulation of the breathing muscles. For comparison: In obstructive apneas are caused by blocked airways that shut off the air although the breathing Stimulus is working.
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: %central/totalapnea
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
%central/totalapnea | 44.6 (28.9) | 46.5 (30.0)

25. Secondary Outcome: Central AHI/Total AHI at Baseline
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: Central/totalAHI%
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
Central/totalAHI% | 80.8 (15.5) | 81.8 (15.7)

26. Secondary Outcome: Oxygen Desaturation Index (ODI) at Baseline
Description: Number of oxygen desaturations per hour at baseline
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
events/hour | 32.1 (17.7) | 32.8 (19.0)

27. Secondary Outcome: Oxygen Saturation Baseline
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: %total hemoglobine
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
%total hemoglobine | 92.8 (2.3) | 92.8 (2.5)

28. Secondary Outcome: Time With Oxygen Saturation Below 90%
Time Frame: 1 x at baseline
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 666 | 659
min | 50.5 (68.2) | 55.7 (73.9)

29. Secondary Outcome: Time Until Unplanned Hospitalisation/Prolongation of Hospitalisation for Cardiovascular Cause or Cardiovascular Death/ Time Frame
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected.
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Percent of Follow up Days Which Patient Survives and is Not Hospitalized/Hospital Stay is Not Prolonged for Cardiovascular Cause
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Changes in NYHA Classification as Compared to Baseline
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Changes in QoL (Minnesota) as Compared to Baseline
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Changes in Renal Function (Based on Serum Creatinine) as Compared to Baseline
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Changes in Six Minute Walking Distance (6MWD) as Compared to Baseline
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Changes of AHI and Oxygen Desaturation Index Compared to Baseline
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: AHI Below 10 Per Hour at Twelve Months and ODI Below 5 Per Hour at Twelve Months
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Atrial Fibrillation at Follow-up Visits
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Number and Cost of Hospitalisations (With Tariff/DRG, Diagnoses and Procedures for Calculating DRG or Length of Stay and Level of Care Provided)
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Difference in Utilities / QoL (Minnesota and EQ5D) Compared to Control Arm
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Difference in Cost of Resources Consumed
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Incremental Cost-efficacy Ratio
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Incremental Cost-utility Ratio
Time Frame: the last follow up or at the last available observation within FU, assessed for up to 70 weeks
Population: Data have not been collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 232/666 | 193/659
Serious Adverse Events (participants affected / at risk) | 482/666 | 465/659
Other Adverse Events (participants affected / at risk) | 0/666 | 0/659
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=666) | Control Group (N=659)
Cardiovascular death (Cardiac disorders) | 199 (199) | 158 (158)
Primary end point (General disorders) | 360 (360) | 335 (335) — First event of death from any cause, lifesaving cardiovascular intervention, unplanned hospitalization for worsening chronic heart failure
Firt secondary endpoint (Cardiac disorders) | 345 (345) | 317 (317) — First Event of cardiovascular death, lifesaving cardiovascular Intervention, unplanned hospitalization for worsening chronic heart failure
Second secondary endpoint (General disorders) | 482 (482) | 465 (465) — First event of death from any cause, lifesaving cardiovascular intervention, unplanned hospitalization for any cause
Hospitalization for any cause (General disorders) | 452 (452) | 448 (448)
Unplanned hospitalization for worsening heart failure (Cardiac disorders) | 287 (287) | 272 (272)
Heart transplantation (Cardiac disorders) | 8 (8) | 12 (12)
Implantation of long-term VentricularAssistDev (Cardiac disorders) | 16 (16) | 10 (10)
Resuscitation (General disorders) | 25 (25) | 19 (19)
Resuscitation for cardiac arrest (Cardiac disorders) | 18 (18) | 16 (16)
Appropriate Shock for ventricular arrhythmia (Cardiac disorders) | 45 (45) | 65 (65)
Noncardiovascular death (General disorders) | 33 (33) | 35 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No